CLINICAL TRIAL: NCT01817985
Title: A Phase 1 Open-Label, Parallel-Group, Single-Dose Study to Evaluate the Pharmacokinetics of GS-5816 in Subjects With Normal Hepatic Function and Moderate or Severe Hepatic Impairment
Brief Title: A Phase 1 Study to Evaluate the Pharmacokinetics of GS-5816 in Subjects With Normal Hepatic Function and Moderate or Severe Hepatic Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-281-0112
Record Dates: First submitted 2013-03-20; First posted 2013-03-26 (Estimated); Last update posted 2013-08-29 (Estimated); Status verified 2013-08

CONDITIONS: Chronic Hepatitis C
Keywords: Hepatitis C (HCV) Infection; Moderate Hepatic Impairment; Severe Hepatic Impairment
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C; Infections | interventions — velpatasvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort 1 (Experimental): (N = 20 Moderately Impaired / Normal Hepatic Function) 100 mg GS-5816.
  Interventions: Drug: GS-5816
- Cohort 2 (Experimental): (N = 20 Severely Impaired / Normal Hepatic Function) up to 100 mg GS-5816.
  Interventions: Drug: GS-5816

INTERVENTIONS:
Drug: GS-5816

SUMMARY:
This is a Phase 1 Open-Label, Parallel-Group, Single-Dose Study to evaluate the Pharmacokinetics of GS-5816 in subjects with normal hepatic function and moderate or severe hepatic impairment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic (> 6 months), hepatic impairment.
* In the opinion of the Investigator, be in good health.

Exclusion Criteria:

* Severe hepatic encephalopathy.
* Prior placement of a portosystemic shunt.
* Hepatorenal or hepatopulmonary syndrome.
* Suspicion of hepatocellular carcinoma.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2013-03; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters of GS-5816 | Up to one year
  The primary outcome measure is the pharmacokinetic parameters of GS-5816 which will include AUClast, AUCinf, and Cmax.

SECONDARY OUTCOMES:
Incidences of adverse events and laboratory abnormalities | Up to one year
  The secondary outcome measure is the number of incidences of adverse events and laboratory abnormalities.

CONTACTS AND LOCATIONS:
Overall Officials: Diana Brainard, M.D., Study Director — Gilead Sciences
Locations (4):
- United States (3):
  - Investigational Site, Miami, Florida
  - Investigational Site, Orlando, Florida
  - Investigational Site, San Antonio, Texas
- Investigational Site, San Juan, Puerto Rico, Puerto Rico